CLINICAL TRIAL: NCT06909565
Title: Evaluation of Inclisiran Versus Placebo for the Prevention of Major Adverse Cardiovascular and Limb Events in Patients Undergoing Percutaneous Coronary Intervention or Peripheral Endovascular Intervention (V-INTERVENTION)
Brief Title: Inclisiran Versus Placebo for the Prevention of Major Adverse Cardiovascular and Limb Events in Patients Undergoing Percutaneous Coronary Intervention or Peripheral Endovascular Intervention
Acronym: V-INTERVENTION
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Colorado Prevention Center (Other); Mount Sinai Hospital, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00116826; CKJX839D1US04R (Other: Novartis Pharmaceuticals Corporation)
Record Dates: First submitted 2025-03-27; First posted 2025-04-03 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-07

CONDITIONS: Percutaneous Coronary Intervention; Peripheral Endovascular Intervention
Keywords: inclisiran; Coronary Artery Disease; hypercholesterolemia; Cardiovascular Disease; Percutaneous Endovascular Intervention; Percutaneous Coronary Intervention; PCSK9
MeSH Terms: conditions — Coronary Artery Disease; Hypercholesterolemia; Cardiovascular Diseases | interventions — ALN-PCS; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Inclisiran Sodium (Active Comparator): Inclisiran sodium 300 mg subcutaneous injection
  Interventions: Drug: Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) in 1.5 mL
- Placebo (Placebo Comparator): Normal saline 1.5 ml subcutaneous injection
  Interventions: Drug: Normal Saline (Placebo)

INTERVENTIONS:
Drug: Inclisiran sodium 300 mg (equivalent to 284 mg inclisiran) in 1.5 mL — 300 mg (equivalent to 284 mg inclisiran) in 1.5 mL subcutaneous injection at Day 0; Day 90; & every 6 months thereafter
  Arms: Inclisiran Sodium
Drug: Normal Saline (Placebo) — Normal saline placebo subcutaneous injection given at Day 0, Day 90; & every 6 months thereafter
  Arms: Placebo

SUMMARY:
V-INTERVENTION will evaluate the effectiveness of inclisiran in preventing major cardiovascular and limb events in patients receiving percutaneous coronary or peripheral arterial revascularization. Inclisiran is a subcutaneous, twice-yearly injection that is FDA-approved as an adjunct with statin therapy and on the market to lower LDL-C in high-risk populations.

DETAILED DESCRIPTION:
CKJX839D1US04R is a pragmatic, randomized, double-blind, parallel group, placebo-controlled, multicenter, event-driven study evaluating inclisiran sodium 300 mg subcutaneous administered on Day 1, Month 3 (Day 90), and every 6 months thereafter in participants presenting for elective or urgent percutaneous coronary or peripheral endovascular intervention (PCI or PVI). At the time of a successful revascularization procedure or up to 14 days following the procedure, participants will be randomized and administered the first dose of inclisiran or corresponding placebo in a 1:1 fashion, stratified by the type of index arterial revascularization procedure, either coronary (i.e., PCI) or lower extremity (i.e., PV).

The enrollment population will be representative of typical patients in the US with atherosclerotic cardiovascular disease, either coronary artery disease (CAD) or peripheral artery disease (PAD), and the trial endpoints are designed to be scientifically relevant and clinically meaningful to patients, clinicians, and other persons involved in the care of cardiovascular patients. The trial is designed to also understand how inclisiran therapy can be implemented in real-world clinical practice settings.

The expected enrollment of the trial is approximately 6,000 participants, randomized in a 1:1 fashion to receive inclisiran or placebo, within 14 days of successful percutaneous coronary or lower extremity peripheral endovascular intervention for symptomatic atherosclerotic cardiovascular disease (ASCVD).

Inclisiran sodium or corresponding placebo will be administered by s.c. injection to participants presenting for percutaneous coronary or peripheral endovascular intervention, in addition to usual care according to their individual medical history. All participants randomized to the treatment arm will receive inclisiran in addition to usual care per their regular physician direction, and those participants randomized to placebo will receive matching placebo, as well as usual care treatment, according to their treating physician.

Study duration is determined by event accrual consistent with the event-driven design, i.e., when approximately 2380 primary composite events have occurred and at least 50% of participants have at least 36 months of follow-up. Assuming 18 months of recruitment at a uniform rate, the last patients enrolled will have about 27 months of follow-up. Therefore, study duration should be approximately 4 years.

The study is event-driven, and thus, all participants will be treated (or followed in the case of permanent discontinuation of study drug) until the End of Study visit. As such, the planned duration of treatment cannot be stipulated for an individual participant. The estimated maximum treatment period for an individual participant is approximately 45 months, and the mean treatment duration is expected to be approximately 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Males or females ≥ 18 years of age
* Within 14 days of a successful percutaneous coronary intervention (PCI) or peripheral endovascular intervention (PVI) for symptomatic CAD or lower extremity PAD
* Patients undergoing planned staged interventions are eligible for randomization only after the last planned intervention

Exclusion Criteria:

* Planned future PCI or PVI
* Current or planned use of an open-label PCSK9 inhibitor during the study
* Any prior treatment with inclisiran
* Active or planned participation in another clinical study involving investigational drugs or devices during the study
* Any serious liver disease, metabolic disease, neoplasm, end-stage kidney disease, or other condition in the opinion of the investigator that would inhibit trial participation or confound trial results
* Any other reason why, in the opinion of the investigator, the participant would not be suitable for study participation including safety considerations and the ability to adhere to protocol activities
* Patients taking prohibited therapies as listed in Section 6.6.3
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Total number of major adverse cardiovascular events (MACE) after coronary or peripheral endovascular revascularization | From randomization to first occurrence of MACE (up to approximately 4 years)
  MACEs include CHD death, non-fatal MI, ischemic stroke, ALI, major (above the ankle) amputation of vascular etiology, clinically driven coronary and limb revascularization.
Total number of major adverse limb events (MALE) after endovascular revascularization | From randomization to first occurrence of MALE (up to approximately 4 years)
  MALEs consist of ALI, major amputation of vascular etiology, clinically driven lower extremity peripheral revascularization.

SECONDARY OUTCOMES:
Number of participants with cardiovascular (CV) death | From randomization to CV death (up to approximately 4 years)
Number of participants with all cause death | From randomization to all cause death (up to approximately 4 years)
Number of participants with venous thromboembolic events (VTE) | From randomization to first VTE (up to approximately 4 years)

CONTACTS AND LOCATIONS:
Overall Officials: Schuyler Jones, MD, Principal Investigator — Duke Clinical Research Institute; Marc Bonaca, MD, Principal Investigator — Colorado Prevention Center; Roxana Mehran, MD, Study Chair — Mt Sinai; Manesh Patel, MD, Study Chair — Duke University
Locations (53):
- United States (53):
  - Advanced Cardiovascular LLC, Alexander City, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Arkansas Cardiology, Little Rock, Arkansas
  - Pacific Oaks Medical Group, Beverly Hills, California
  - Valley Clinical Trials, Covina, California
  - Radin Cardiovascular Medical Group, Inc, Newport Beach, California
  - Valley Clinical Trials, LLC - Flourish Research, Northridge, California
  - The Heart Medical Group, Van Nuys, California
  - Interventional Cardiology Medical Group, West Hills, California
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Pioneer Clinical Studies, Coral Gables, Florida
  - Arrow Clinical Trails, Daytona Beach, Florida
  - Clearwater Cardiovascular and Interventional Consultants- Bardmoor, Largo, Florida
  - Inpatient Research Clinic, LLC, Miami Lakes, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - Charlotte Heart & Vascular Center, PA, Port Charlotte, Florida
  - Clearwater Cardiovascular Consultants, Safety Harbor, Florida
  - Tampa Cardiovascular Interventions and Research, Tampa, Florida
  - Reid Physician Associates, Richmond, Indiana
  - Midwest Heart and Vascular Specialists, Overland Park, Kansas
  - Grace Research, LLC, Bossier City, Louisiana
  - Louisiana Heart Center, Covington, Louisiana
  - Cardiovascular Solutions, LLC, Shreveport, Louisiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - UMH-Sparrow Clinical Research Institute, Lansing, Michigan
  - MyMichigan Medical Center Midland, Midland, Michigan
  - Healthy Heart Cardiology at Rochester Hills (Advanced Cardiology Associates, Rochester Hills, Michigan
  - CHI Health Nebraska Heart, Grand Island, Nebraska
  - CHI Health Nebraska Heart, Lincoln, Nebraska
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Elmer, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Cardiovascular Associates of the Delaware Valley, Sewell, New Jersey
  - Trinity Medical WNY, PC, Buffalo, New York
  - Mount Sinai School of Medicine, New York, New York
  - Richmond University Medical Center, Staten Island, New York
  - Mecklenburg Heart Specialists, Charlotte, North Carolina
  - Duke Cardiology, Morrisville, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Heart House Research Foundation LLC, Springfield, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Capital Area Research LLC, Camp Hill, Pennsylvania
  - WellSpan Heart and Vascular Research, York, Pennsylvania
  - AnMed Health Medical Center, Anderson, South Carolina
  - Apex Research Foundation, LLC, Jackson, Tennessee
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - Amarillo Heart Clinical Research Institute, Inc., Amarillo, Texas
  - Heart Institute of East Texas, Lufkin, Texas
  - TPMG Clinical Research, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navar AM, Shah NP, Shrader P, Thomas LE, Ahmad Z, Allred C, Chamberlain AM, Chrischilles EA, Dhalwani N, Effron MB, Hayek S, Jones LK, Kalich B, Shapiro MD, Wojcik C, Peterson ED. Achievement of LDL-C <55 mg/dL among US adults: Findings from the cvMOBIUS2 registry. Am Heart J. 2025 Jan;279:107-117. doi: 10.1016/j.ahj.2024.06.012. Epub 2024 Jul 6. PMID 38972336
- [Background] Chamberlain AM, Gong Y, Shaw KM, Bian J, Song WL, Linton MF, Fonseca V, Price-Haywood E, Guhl E, King JB, Shah RU, Puro J, Shenkman E, Pawloski PA, Margolis KL, Hernandez AF, Cooper-DeHoff RM. PCSK9 Inhibitor Use in the Real World: Data From the National Patient-Centered Research Network. J Am Heart Assoc. 2019 May 7;8(9):e011246. doi: 10.1161/JAHA.118.011246. PMID 31020929